CLINICAL TRIAL: NCT02746718
Title: Frequency of Pompe's Disease and Neuromuscular Etiologies in Patients With Restrictive Respiratory Failure Associated With Signs of Muscle Weakness
Acronym: POPS3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-PP-13
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2018-03

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restrictive Respiratory Failure (Other): A CPK dosage, muscular questionnaires and a Pompe Disease test are practiced on patient with Restrictive Respiratory Failure without etiology
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample for CPK dosage and pompe disease test

SUMMARY:
A breach of respiratory function may be one of the elements more or less early or predominant clinical picture of neuromuscular diseases. It is considered that the obstructive syndromes represent 64% and restrictive or mixed syndromes 36% of chronic respiratory insufficiency, approximately 7% due to a neuromuscular disease. The frequency and type of impairment are dependent on the underlying pathology.

The neuromuscular restrictive respiratory failure (IRR) remains partially unknown pulmonologists, especially because the signs of muscle weakness are sometimes difficult to detect. However, respiratory diseases are a major concern in neuromuscular diseases because they can have an impact both on sleep (not sleep, ...) on the daily activities (breathlessness on exertion, dyspnea) and thereby alter the quality of life of patients. Moreover, they represent a significant morbidity and mortality factor. Chest tightness may in some cases reveal the disease and thus constitute the chief complaint of a patient with a neuromuscular disease. In late-onset Pompe disease, lung disease is the predominant clinical symptoms in about 30% of patients.

An algorithm was developed to guide practitioners and help them in their diagnostic approach to the cause of the IRR (diagnostic algorithm ATS / ERS 2005). However, this algorithm does not allow precise identification of the neuromuscular causes.

At the patient level, this can have an impact by extending the time before placing a diagnosis. In Pompe disease, the average time to diagnosis reached 7.9 years. However, there are for this disease a simple and rapid diagnostic test. Therefore, a greater awareness of practitioners with regard to the particular Pompe disease and neuromuscular diseases in general may be beneficial to patients.

This study aims to:

i) awareness pulmonologists to the possibility of neuromuscular an IRR.

ii) characterize the frequency of neuromuscular origin of IRR in a broad population of patients with concomitant signs muscle weakness.

iii) reduce the time to diagnosis by directing patients to neuromuscular reference center early.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a CV <80% of predicted and / or <LIN
* Presence spirometry a report Tiffeneau (FEV / CV) equal to or higher than normal
* Signature of informed consent
* Men and women age ≥ 18 years
* Production of a medical examination
* Affiliated to social security

Exclusion Criteria:

* restrictive breath traumatic
* restrictive respiratory failure associated with parenchymal disorder, whether localized or diffuse
* known neuromuscular disease associated with a restrictive lung disease
* Patient under guardianship, curatorship, protected by law
* Inability to cooperate
* Morbid obesity with a BMI ≥40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Number of new cases of Pompe disease diagnosed by a positive DBS | At the inclusion
  Number of new cases of Pompe disease diagnosed by a positive DBS in patients with unexplained restriction pulmonaires.ries volumes, the patient is adressed to a specialist to dertermine etilogy of the muscular disease.

SECONDARY OUTCOMES:
Number of new cases and etiologies of neuromuscular diseases diagnosed in patients with unexplained restriction of lung volumes | at 6 month
  If a patient have an high CPK rate or a blotter test positive for Pompe disease or a suspicion of muscular disease with the muscular questionnaires, the patient is addressed to a specialist to determine etiology of the muscular disease.
Frequency and description of neurological symptoms associated with neuromuscular diseases to respiratory revelation | at 6 month
  If a patient have an high CPK rate or a suspicion of muscular disease with the muscular questionnaires, the patient is addressed to a specialist to determine etiology of the muscular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Sacconi, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (21):
- France (21):
  - CHU d'Angers, Angers
  - Centre hospitalier d'Argenteuil, Argenteuil
  - CHU de Brest, Brest
  - CH d'Escartons, Briançon
  - CH de Cannes, Cannes
  - CHI de Créteil, Créteil
  - CHU le Bocage, Dijon
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - Cabinet Dr Pereira-Cortese, Nice
  - CHU de Nice, Nice
  - GH Pitié Salpêtrière, Paris
  - Hôpital Raymond Poincaré, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Tenon, Paris
  - Polyclinique les Bleuets, Reims
  - CHU de Rouen, Rouen
  - CHU de St Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours
  - Clinique Saint Joseph, Trélazé

IPD SHARING:
Plan to Share IPD: No